CLINICAL TRIAL: NCT05128981
Title: Internet-delivered Cognitive Behavioral Therapy Following Myocardial Infarction
Acronym: MI-CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Josefin Särnholm, PhD, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBT-MI
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Myocardial Infarction; Cardiac Anxiety; CBT; Exposure
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MI-CBT via the Internet (Other): The MI-specific CBT will consist of 8 modules delivered via the Internet with home assignments that can be reviewed and reported in the research groups secure platform.
  Interventions: Behavioral: MI-CBT

INTERVENTIONS:
Behavioral: MI-CBT — Education of MI and common reactions, Interoceptive exposure, Exposure in-vivo, Behavioral activation, Relapse prevention

SUMMARY:
Myocardial infarction (MI) is one of the leading cause s of health loss globally, representing a large proportion of general disability. Anxiety and depression occur in 20-30 percent of patients following MI and have been identified as risk factors for recurrent adverse cardiac event. The purpose of our this study is to develop and evaluate a disease specific cognitive behavioral therapy (C BT) protocol to reduce cardia anxiety, depression, increase physical inactivity and quality of life (Q oL) in patients following MI

DETAILED DESCRIPTION:
The study will include 30 patients. The MI-specific CBT lasts for 8 weeks and is therapist guided and delivered via internet via a secure digital platform by licensed psychologists expertise in CBT for cardiac disease or final year psychologist under supervision. During treatment, the psychologists will have direct access to a cardiologist assigned to the project and treatments are conducted in close interdisciplinary collaboration to ensure patient safety

ELIGIBILITY:
Inclusion Criteria:

( - )MI ≥ 6 months before assessment ( - )Age 18-75 years endorsed cardiac anxiety that leads to significant distress or interferes with daily life (Cardiac Anxiety Questionnaire (CAQ); score ≥20) ( - ) On optimal medical treatment ( - )Able to read and write in Swedish.

Exclusion Criteria:

( - ) heart failure with severe systolic dysfunction (ejection fraction ≤ 35%) ( - ) significant valvular disease ( - ) planned coronary artery bypass surgery or other invasive therapy ( - ) other severe medical illness ( - )any medical restriction to physical exercise ( - )severe psychiatric disorder, severe depression, or risk of suicide ( - )alcohol dependency

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
12-Item Short-Form Health Survey (SF-12) | Baseline
  General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life.
  General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life.
  General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life.
12-Item Short-Form Health Survey (SF-12) | 2 months from baseline
  General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life.
  General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life.
  General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life.
12-Item Short-Form Health Survey (SF-12) | 8 months from baseline
  General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life.
  General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life.
  General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life.

SECONDARY OUTCOMES:
Cardiac anxiety questionnaire | Baseline
  Measure of cardiac anxiety, fear, avoidance and attention. The score ranges between 0 and 72, with a greater score indicating elevated cardiac anxiety.
Cardiac anxiety questionnaire | 2 months from baseline
  Measure of cardiac anxiety, fear, avoidance and attention. The score ranges between 0 and 72, with a greater score indicating elevated cardiac anxiety.
Cardiac anxiety questionnaire | 8 months from baseline
  Measure of cardiac anxiety, fear, avoidance and attention. The score ranges between 0 and 72, with a greater score indicating elevated cardiac anxiety.
Body Sensation Questionnaire | Baseline
  Fear of bodily symptoms, score ranging from 0 to 72 . Higher scores indicate more fear of body sensations.
  Fear of bodily symptoms, score ranging from 0 to 72 . Higher scores indicate more fear of body sensations.
  Fear of bodily symptoms, score ranging from 0 to 72 . Higher scores indicate more fear of body sensations.
Body Sensation Questionnaire | 2 months from baseline
  Fear of bodily symptoms, score ranging from 0 to 72 . Higher scores indicate more fear of body sensations.
  Fear of bodily symptoms, score ranging from 0 to 72 . Higher scores indicate more fear of body sensations.
  Fear of bodily symptoms, score ranging from 0 to 72 . Higher scores indicate more fear of body sensations.
Body Sensation Questionnaire | 8 months from baseline
  Fear of bodily symptoms, score ranging from 0 to 72 . Higher scores indicate more fear of body sensations.
  Fear of bodily symptoms, score ranging from 0 to 72 . Higher scores indicate more fear of body sensations.
  Fear of bodily symptoms, score ranging from 0 to 72 . Higher scores indicate more fear of body sensations.
Patient Health Questionnaire-9 | Baseline
  Measure of depression, score ranging 0 to 27 with a higher score indicating higher level of depression
Patient Health Questionnaire-9 | 2 months from baseline
  Measure of depression, score ranging 0 to 27 with a higher score indicating higher level of depression
Patient Health Questionnaire-9 | 8 months from baseline
  Measure of depression, score ranging 0 to 27 with a higher score indicating higher level of depression
Generalized Anxiety Disorder 7-item | Baseline
  General anxiety, score ranging from 0-21, with a higher score indicating more anxiety and worry.
Generalized Anxiety Disorder 7-item | 2 months from baseline
  General anxiety, score ranging from 0-21, with a higher score indicating more anxiety and worry.
Generalized Anxiety Disorder 7-item | 8 months from baseline
  General anxiety, score ranging from 0-21, with a higher score indicating more anxiety and worry.
The Godin Leisure-time Exercise | Baseline
  Level of physical activity. The participant rate numbers of time per week that they engage in physical activity. The numb ers are the categorized in to low, moderate, and high levels of physical activity.
The Godin Leisure-time Exercise | 2 months from baseline
  Level of physical activity. The participant rate numbers of time per week that they engage in physical activity. The numb ers are the categorized in to low, moderate, and high levels of physical activity.
The Godin Leisure-time Exercise | 8 months from baseline
  Level of physical activity. The participant rate numbers of time per week that they engage in physical activity. The numb ers are the categorized in to low, moderate, and high levels of physical activity.
Tampas Scale for Kinesophobia-Heart version | Baseline
  Fear of physical activity. The total score varies between 17 and 68, with higher values indicating more severe kinesiophobia.
Tampas Scale for Kinesophobia-Heart version | 2 months from baseline
  Fear of physical activity. The total score varies between 17 and 68, with higher values indicating more severe kinesiophobia.
Tampas Scale for Kinesophobia-Heart version | 8 months from baseline
  Fear of physical activity. The total score varies between 17 and 68, with higher values indicating more severe kinesiophobia.
Client satisfaction Questionnaire | Baseline
  Treatment satisfaction, score ranging from 0 to 32, with a higher score indication more satisfaction with the treatment.
Client satisfaction Questionnaire | 2 months from baseline
  Treatment satisfaction, score ranging from 0 to 32, with a higher score indication more satisfaction with the treatment.
Adverse events | 2 months from treatment
  Potential adverse reactions to the treatment. Participants will be asked to report and rate the short- and long term discomfort of the adverse event on a scale from 0 ('did not affect me at all') and 3 ('affected me very negatively').
Adverse events | 8 months from treatment
  Potential adverse reactions to the treatment. Participants will be asked to report and rate the short- and long term discomfort of the adverse event on a scale from 0 ('did not affect me at all') and 3 ('affected me very negatively').
Symptom Checklist (SCL) | Baseline
  Measures frequency and severity of 16 cardiac-related symptoms. Scoring range from 0 to 64 for frequency with a greater score indicating more frequent symptoms, and from range from 0 to 48 for severity, with a greater score indicating more severe symptoms
Symptom Checklist (SCL) | 2 months from baseline
  Measures frequency and severity of 16 cardiac-related symptoms. Scoring range from 0 to 64 for frequency with a greater score indicating more frequent symptoms, and from range from 0 to 48 for severity, with a greater score indicating more severe symptoms
Symptom Checklist (SCL) | 8 months from baseline
  Measures frequency and severity of 16 cardiac-related symptoms. Scoring range from 0 to 64 for frequency with a greater score indicating more frequent symptoms, and from range from 0 to 48 for severity, with a greater score indicating more severe symptoms
Perceived stress scale (4-item version) | Baseline
  Stress reactivity. A greater score indicate more perceived stress.
Perceived stress scale (4-item version) | 2 months from Baseline
  Stress reactivity. A greater score indicate more perceived stress.
Perceived stress scale (4-item version) | 8 months from Baseline
  Stress reactivity. A greater score indicate more perceived stress.
Insomnia Severity Index | Baseline
  Measurement of sleep
Insomnia Severity Index | 2 months from Baseline
  Measure of insomnia, score ranging from 0-20, with a higher score indicating more severe insomnia
Insomnia Severity Index | 8 months from Baseline
  Measure of insomnia, score ranging from 0-20, with a higher score indicating more severe insomnia
The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) | Baseline
  Measure of post traumatic stress, score ranging from 0-80, with a higher score indicating more post traumatic stress.
The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) | 2 months from Baseline
  Measure of post traumatic stress, score ranging from 0-80, with a higher score indicating more post traumatic stress.
The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) | 8 months from Baseline
  Measure of post traumatic stress, score ranging from 0-80, with a higher score indicating more post traumatic stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No